CLINICAL TRIAL: NCT05461833
Title: Fecal Microbiota Transplantation in Patients With Post-infection Irritable Bowel Syndrome: a Randomized, Clinical Trial
Brief Title: FMT for Post-infectious IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Ukrainian Research and Practical Centre of Endocrine Surgery, Transplantation of Endocrine Organs and Tissues of the Ministry of Health of Ukraine (Unknown)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-PI-IBS
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; fecal microbiota transplantation; postinfectious irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation; octylonium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal transplantation group (Experimental): Fecal transplantation of frozen prepared feces from healthy donor. Application by colonoscope in proximal half of colon.
  Interventions: Biological: Fecal transplantation
- Standard-care group (Active Comparator): FODMAP diet, Otilonium Bromide, oral, (40mg, 1 tablet TID) and a multi-strain probiotic, oral, (1 capsule BID)
  Interventions: Drug: OTILONII BROMIDUM; Dietary Supplement: multi-strain probiotic

INTERVENTIONS:
Biological: Fecal transplantation — Preparation of flesh feces by blending in 0.9 % saline and crude filtering. The solution is applied in proximal colon of IBS patient by colonoscopy after standard bowel preparation.
  Other Names: Fecal microbial transplantation
  Arms: Fecal transplantation group
Drug: OTILONII BROMIDUM — OTILONII BROMIDUM , oral, 40 mg TID, 1 months of treatment
  Other Names: Spasmomen®
  Arms: Standard-care group
Dietary Supplement: multi-strain probiotic — multi-strain probiotic, oral, 1 capsule BID for 1 month
  Arms: Standard-care group

SUMMARY:
Considering that PI-IBS is brought on by infection and gut microbiota may be associated with the onset of symptoms, the modification of altered gut microbiota with nonabsorbable antibiotics such as rifaximin-α or probiotics is often employed as first-stage treatment. Research in recent years has also shown the potential benefits of fecal microbiota transplantation (FMT) for IBS, which is the replacement of a sick recipient's gut microbiota with fecal material from a healthy donor. Even though the only officially approved indication for FMT at this time is recurrent Clostridium difficile infection, the effectiveness of FMT is nevertheless being studied for the treatment of other gastrointestinal and non-gastrointestinal pathologies including IBS. To date, several controlled and uncontrolled studies have been conducted to study the effectiveness of FMT for IBS, and most of them have demonstrated positive results. The investigators have not come across studies devoted to the study of the effectiveness of FMT in patients with PI-IBS in the available literature. So, the aim of the current study was to conduct single-centre, randomized clinical trial to assess the safety, clinical and microbiological efficacy of FMT in patients with PI-IBS.

ELIGIBILITY:
Inclusion Criteria

* age 18-65 years
* PI-IBS diagnosis in accordance with the Rome IV criteria
* moderate-severe disease activity (as determined by an IBS-Symptom Severity Score ≥175)
* normal appearing colon on colonoscopy with biopsy that did not reveal pathology
* signed inform consent.

Exclusion Criteria:

* systemic disease, immunodeficiency, or previous treatment with immunomodulators;
* pregnant or breastfeeding;
* previous surgery on the abdominal cavity, with the exception of appendectomy, cholecystectomy, caesarean section and hysterectomy;
* severe current disease (hepatic, renal, respiratory, or cardiovascular);
* probiotic or antibiotic use within 8 weeks prior to study initiation;
* any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Irritable bowel syndrome severity scoring system (IBS-SSS) | at 0, 2, 4 and 12 weeks
  This questionnaire contains five questions, each with a maximum score of 100 using a visual analog scale. Total scores between 75 and 175 were considered indicative of mild IBS severity, 175-300 were moderate, and >300 were severe.
assesment of response rate | at 12 weeks
  response rate was assessed as decrease of ≥ 50 points on the IBS-SSS

SECONDARY OUTCOMES:
Change in BS Quality of Life Scale (IBS-QoL) | at 0, 2, 4 and 12 weeks
  This questionnaire contains 34 items concerning the physical and psychological functioning of IBS patients in 8 domains: dysphoria, activity interference, body image, health concerns, food avoidance, social reactions, sexual function and impact on relationships.
Change in Fatigue Assessment Scale (FAS) | at 0, 2, 4 and 12 weeks
  The questionnaire comprises 10 questions with 5-point-scale answers varying from never to always. Five of these questions measured physical fatigue and the other five measured mental fatigue.
Bacteriology measured in the stool flora by specialized non-culture techniques | at 0 and 1 months
  The percentage of patients in each group were evaluated and characterized by a decrease below the normal content of symbiotic bacteria Bifidobacterium (less than 107 CFU / g), lactobacilli (less than 107 CFU / d), E.coli with normal properties (less than 106 CFU / d) and increase in content E.coli with altered properties (more than 106 CFU / g), pathogenic enterobacteria (not normally detected) and fungi of the genus Candida (more than 104 CFU / d)
Microbiome profile change | at 0 and 1 months
  Characterization of fecal microbiome by metagenomic analysis before and after intervention Characterization of fecal microbiome by metagenomic analysis before and after intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - Bogomolets National Medical University, Kyiv
  - Ukrainian Research and Practical Centre of Endocrine Surgery, Transplantation of Endocrine Organs and Tissues of the Ministry of Health of Ukraine, Kyiv

IPD SHARING:
Plan to Share IPD: No